CLINICAL TRIAL: NCT02343861
Title: The Effectiveness of Tailored Messages on the Usage of Emollient in Patients With Atopic Dermatitis: A Pilot Study
Brief Title: The Effectiveness of Tailored Messages on the Usage of Emollient in Patients With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Sun Yoon, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-2014-154
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Dermatitis, Atopic
Keywords: Behavioral Research; Emollients
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored leaflet group (Active Comparator): Participants (parents of children with atopic dermatitis) receive a tailored leaflet about the detailed amount of emollients as well as general information about use of emollients.
  Interventions: Behavioral: Tailored leaflet group
- Control group (Placebo Comparator): Participants (parents of children with atopic dermatitis) receive general information about use of emollients only.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Tailored leaflet group — Parents in intervention group will receive an patient education leaflet and watch an educational video about lifestyle recommendations, and the use of emollients. In addition to general information, parents in intervention group will also receive the tailored leaflet including the estimated amount of emollients based on the body surface area.
  Other Names: Tailored leaflet about the adequate use of emollient
  Arms: Tailored leaflet group
Behavioral: Control group — Participants (parents of children with atopic dermatitis) in control group will receive an patient education leaflet and watch an educational video about lifestyle recommendations, and the use of emollients.
  Arms: Control group

SUMMARY:
Atopic dermatitis is the most common chronic inflammatory skin disease in children and severely affects quality of life (QoL) of patients and their parents. The application of topical medications and emollient is the mainstay of the treatment, but complexity of the treatment and lack of self-care knowledge cause poor adherence, leading to therapeutic failure. Adequate education about the chronic disease and its treatment was known to improve the treatment adherence. There are a variety forms like generalized information leaflets and video clips for imparting information to patients and individualized tailoring education was considered more effective way to improve patients' adherence. The aim of this study is to determine the efficacy of tailored education in dermatology area, especially the emollient usage in patients with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* A parent of 0-5 year old children with mild to moderate atopic dermatitis
* 20 years of age or older
* Apply emollient for themselves to their children with atopic dermatitis

Exclusion Criteria:

* Parents of children with severe atopic dermatitis or showing signs of acute infection (Oozing, vesicles, edema, redness or pain)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change of the weekly amount of emollient used | Two weeks
  Parents of patients are asked to bring the emollients to each visit at which time the emollients are weighed.

SECONDARY OUTCOMES:
Average daily number of emollient usage | Two weeks
Average daily number of topical medication (other than emollient) usage | Two weeks
Investigator's Global Assessment (IGA) | Two weeks
  At each visit, disease severity will be assessed using the Investigator's Global Assessment (IGA).
Eczema Area and Severity Index (EASI) | Two weeks
  At each visit, disease severity will be assessed using the Eczema Area and Severity Index (EASI).

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Sun Yoon, MD, PhD, Study Director — Department of Dermatology, Seoul National University Boramae Hospital
Locations (1):
- Department of Dermatology, Seoul National University Boramae Hospital, Seoul, South Korea

REFERENCES:
- [Result] Park GY, Park HS, Cho S, Yoon HS. The Effectiveness of Tailored Education on the Usage of Moisturizers in Atopic Dermatitis: A Pilot Study. Ann Dermatol. 2017 Jun;29(3):360-362. doi: 10.5021/ad.2017.29.3.360. Epub 2017 May 11. No abstract available. PMID 28566920